CLINICAL TRIAL: NCT02404532
Title: OSMITTER 316-13-206B Substudy: A Substudy to Measure the Accuracy of Ingestible Event Marker (IEM) Detection by the Medical Information Device #1 (MIND1) System and Determine the Latency Period
Brief Title: Substudy 'B' of the Accuracy of Ingestible Event Marker (IEM) Detection by the Medical Information Device #1 (MIND1)
Acronym: OSMITTER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 316-13-206B
Record Dates: First submitted 2015-03-05; First posted 2015-03-31 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Device Latency
Keywords: OPC-14597 Digital; Aripiprazole; Medical Information Device #1 System (MIND1); Ingestible Event Marker

ARMS (1):
- 1 (Experimental)
  Interventions: Device: MIND1 System

INTERVENTIONS:
Device: MIND1 System — Following placement of the Patch by clinic staff, subjects will ingest one placebo-embedded IEM tablet approximately every other hour, for a total of 4 ingestions. Subjects may eat as they wish over the course of the day. Placebo-embedded IEM tablets are being tested to measure the accuracy of IEM detection by the MIND1 system. Clinic staff will record the time of each ingestion of an IEM. Clinic staff will check the compatible computing device (eg, smartphone) at 30-minute intervals for the presence of a timeline ingestion tile and will record the time it is detected by the MIND1 System compatible computing device (eg, smartphone).

SUMMARY:
The purpose of this study is to determine the accuracy of IEM detection by the MIND1 System by completing a series of Patch applications and IEM ingestions in the clinic.

DETAILED DESCRIPTION:
The OSMITTER study protocol is designed as a master protocol governing multiple substudies for the rapid assessment of candidate subcomponents for the MIND1 System. This substudy is being conducted to determine the accuracy of IEM detection by the MIND1 System by completing a series of Patch applications and IEM ingestions in the clinic. Following placement of the Patch by clinic staff, subjects will ingest one placebo-embedded IEM tablet approximately every other hour, for a total of 4 ingestions.

Placebo-embedded IEM tablets are being tested to measure the accuracy of IEM detection by the MIND1 system. Approximately 30 healthy volunteer subjects will be enrolled in the substudy. The duration of this substudy from Visit 1 (Day 1) to safety follow-up will be approximately 1 week, of which approximately 1 day will be allotted for active subject participation, plus a 1-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or healthy non-pregnant females 18 to 65 years of age at the time of informed consent who are willing to either practice abstinence or 2 barrier methods of birth control or 1 barrier method and an oral contraceptive method.
* Subject must be in good general health (not suffering from a serious chronic mental or physical disorder that has required or may in the near future require urgent medical care).
* Body mass index between 19 to 32 kg/m2 (inclusive).

Exclusion Criteria:

* Subject with a history of skin sensitivity to adhesive medical tape or metals.
* Subject with a history or evidence of a medical condition that would expose him or her to an undue risk of a significant adverse event (AE) or interfere with assessments of safety during the course of the trial.
* Subject has received any investigational product within the last 30 days.
* Subject has a current history of drug or alcohol dependence that meets Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria.
* Subject has the presence of cognitive impairment.
* Subject currently taking antipsychotic medication.
* Subject with a terminal illness.
* Subject with a history of chronic dermatitis.
* Subject with a history of gastrointestinal surgery that could impair absorption.
* Female subject who is breastfeeding and/or who has a positive serum pregnancy test result prior to receiving trial medications.
* Sexually active women of childbearing potential (WOCBP) who will not commit to using 2 forms of approved birth control methods or who will not remain abstinent during this trial and for 30 days following the last dose of trial medication.
* Sexually active males who will not commit to using 2 of the approved birth control methods or who will not remain abstinent for the duration of the trial and for 90 days following the last dose of trial medication.
* No permanent physical residence.
* A diastolic blood pressure reading >95 mm Hg or symptomatic hypotension.
* Any subject who, in the opinion of the investigator, should not participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Peters-Strickland, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (1):
- Walnut Creek, California, United States

REFERENCES:
- [Derived] Jan M, Coppin-Renz A, West R, Gallo CL, Cochran JM, Heumen EV, Fahmy M, Reuteman-Fowler JC. Safety Evaluation in Iterative Development of Wearable Patches for Aripiprazole Tablets With Sensor: Pooled Analysis of Clinical Trials. JMIR Form Res. 2023 Dec 12;7:e44768. doi: 10.2196/44768. PMID 38085556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This sub-study was conducted on 29 healthy male and female participants at a single site (clinic) in United States (US). All enrolled participants received study treatment for 1 day (Visit 1), plus a 1-week (7 [+1] days after the last trial visit) safety follow-up period (via phone call).
Pre-assignment Details: A screening period of 14 days included various procedures such as informed consent form signing, urine pregnancy test, study eligibility review, vital signs measurement, medical history, concomitant medication, baseline & demographic data collection, physical measurement, drugs of abuse test & any adverse events (AEs) assessments.
Groups:
- MIND1 System IEM Detection (All Enrolled Participants): On Day 1, for all enrolled participants, a single adhesive patch (paired with the compatible computing device [eg, smart phone] app) was placed on torso (just above the left costal margin, anywhere from the xyphoid to the left mid-axillary line) before the ingestion of the first placebo-embedded ingestible event marker (IEM) tablet. All participants ingested one placebo-embedded IEM tablet approximately every other hour, for a total of 4 ingestions (hours 0, 2, 4, and 6). Placebo-embedded IEM tablets were tested to measure the accuracy of IEM detection by the medical information device #1 (MIND1) system. Clinic staff recorded the time of each ingestion of an IEM. Clinic staff checked the compatible computing device (eg, smart phone) at 30-minute intervals for the presence of a timeline ingestion tile and recorded the time it was detected by the MIND1 system compatible computing device (eg, smart phone).
Period: Overall Study
Arm/Group | MIND1 System IEM Detection (All Enrolled Participants)
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The enrolled sample included all participants who signed an informed consent form and entered the trial. The Intent-to-Treat (ITT) sample included all participants who ingested at least 1 dose of placebo + IEM, regardless of whether or not ingestion was detected successfully.
Groups:
- MIND1 System IEM Detection (All Enrolled Participants): On Day 1, for all enrolled participants, a single adhesive patch (paired with the compatible computing device [eg, smartphone] app) was placed on torso (just above the left costal margin, anywhere from the xyphoid to the left mid-axillary line) before the ingestion of the first placebo-embedded IEM tablet. All participants ingested one placebo-embedded IEM tablet approximately every other hour, for a total of 4 ingestions (hours 0, 2, 4, and 6). Placebo-embedded IEM tablets were tested to measure the accuracy of IEM detection by MIND1 system. Clinic staff recorded the time of each ingestion of an IEM. Clinic staff checked the compatible computing device (eg, smart phone) at 30-minute intervals for the presence of a timeline ingestion tile and recorded the time it was detected by the MIND1 system compatible computing device (eg, smartphone).
Arm/Group | MIND1 System IEM Detection (All Enrolled Participants)
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Placebo-embedded IEM Detection by the MIND1 System Measured by the Percentage of Participants With IEM Detection Reported for Each of the 4 Time Points
Description: All participants ingested one placebo-embedded IEM tablet approximately every other hour, for a total of 4 ingestions (hours 0, 2, 4, and 6). The time of each ingestion of an IEM was recorded. The compatible computing device (eg, smartphone) was checked at 30-minute intervals for the presence of a timeline ingestion tile and the time was recorded. To measure the accuracy of IEM detection by the MIND1 System using the placebo + IEM by the proportion of participants with IEM detection reported for each of the 4 time points.
Time Frame: Day 1 Visit, at hours 0, 2, 4, 6
Population: ITT sample included all participants who had ingested at least 1 dose of placebo-embedded IEM, regardless of whether or not ingestion was detected successfully.
Measure: Count of Participants; unit: Participants
Groups:
- MIND1 System IEM Detection (All Enrolled Participants): On Day 1, for all enrolled participants, a single adhesive patch (paired with the compatible computing device [eg, smartphone] application) was placed on torso (just above the left costal margin, anywhere from the xyphoid to the left mid-axillary line) before the ingestion of the first placebo-embedded IEM tablet. All participants ingested one placebo-embedded IEM tablet approximately every other hour, for a total of 4 ingestions (hours 0, 2, 4, and 6). Placebo-embedded IEM tablets were tested to measure the accuracy of IEM detection by MIND1 system. Clinic staff recorded the time of each ingestion of an IEM. Clinic staff checked the compatible computing device (eg, smartphone) at 30-minute intervals for the presence of a timeline ingestion tile and recorded the time that was detected by the MIND1 system compatible computing device (eg, smartphone).
Arm/Group | MIND1 System IEM Detection (All Enrolled Participants)
Number analyzed (Participants) | 29
Participants
  Hour 0 | 28
  Hour 2 | 27
  Hour 4 | 28
  Hour 6 | 29

2. Primary Outcome: Latency Period Between the Clinical Site-reported Ingestion Time and the Signal Detection of the Ingestion Event by the Patch
Description: All participants ingested one placebo-embedded IEM tablet approximately every other hour, for a total of 4 ingestions (hours 0, 2, 4, and 6). The time of each ingestion of an IEM was recorded. The compatible computing device (eg, smartphone) was checked at 30-minute intervals for the presence of a timeline ingestion tile and the time was recorded. To evaluate the latency period between site-reported ingestion time and detection of the ingestion event by the patch which displayed on the MIND1 System compatible computing device (eg, smartphone) as a timeline.
Time Frame: Day 1 Visit at 0, 2, 4 and 6 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | MIND1 System IEM Detection (All Enrolled Participants)
Number analyzed (Participants) | 29
Minutes
  Hour 0: number analyzed (Participants) | 28
  Hour 0 | 1.2 (0.8)
  Hour 2: number analyzed (Participants) | 27
  Hour 2 | 1.3 (1.0)
  Hour 4: number analyzed (Participants) | 28
  Hour 4 | 1.1 (1.3)
  Hour 6 | 1.3 (0.9)

3. Secondary Outcome: The Latency Period Between the Patch Detection of an Ingestion Event (eg, the Acquisition Time Stamp) and the Detection of the Ingestion Event in the Otsuka Cloud Server (eg, Server Time Stamp).
Description: All participants ingested one placebo-embedded IEM tablet approximately every other hour, for a total of 4 ingestions (hours 0, 2, 4, and 6). The time of each ingestion of an IEM was recorded. The compatible computing device (eg, smartphone) was checked at 30-minute intervals for the presence of a timeline ingestion tile and the time was recorded. To measure the latency period between the patch detection of an ingestion event and the detection of the ingestion event on the Otsuka Cloud Server which displayed on the MIND1 System compatible computing device (eg, smartphone) as a timeline ingestion tile after each scheduled ingestion event. The various information transmissions measured were patch Acquisition of IEM to Medical Device Data Systems (MDDS), MDDS to Otsuka software application registration, Otsuka software application registration to Cloud Server and patch Acquisition of IEM to Cloud Server
Time Frame: Day 1 Visit at 0, 2, 4 and 6 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Patch Acquisition of IEM to MDDS: The information transmission - Patch Acquisition of IEM to MDDS was measured at all four time points (Hour 0, 2, 4 and 6)
- MDDS to Otsuka Software Application Registration: The information transmission - MDDS to Otsuka software application registration was measured at all four time points (Hour 0, 2, 4 and 6)
- Otsuka Software Application Registration to Cloud Server: The information transmission - Otsuka software application registration to Cloud Server was measured at all four time points (Hour 0, 2, 4 and 6)
- Patch Acquisition of IEM to Cloud Server: The information transmission - Patch acquisition of IEM to Cloud Server was measures at all four time points (Hour 0, 2, 4 and 6)
Arm/Group | Patch Acquisition of IEM to MDDS | MDDS to Otsuka Software Application Registration | Otsuka Software Application Registration to Cloud Server | Patch Acquisition of IEM to Cloud Server
Number analyzed (Participants) | 29 | 29 | 29 | 29
Minutes
  Hour 0: number analyzed (Participants) | 28 | 28 | 28 | 28
  Hour 0 | 5.59 (23.07) | 1.85 (6.38) | 0.01 (0.01) | 7.46 (23.67)
  Hour 2: number analyzed (Participants) | 26 | 26 | 26 | 26
  Hour 2 | 9.74 (21.16) | 0.52 (0.70) | 0.02 (0.01) | 10.28 (20.93)
  Hour 4: number analyzed (Participants) | 27 | 27 | 27 | 27
  Hour 4 | 3.58 (7.84) | 2.62 (7.48) | 0.01 (0.01) | 6.21 (10.36)
  Hour 6 | 4.00 (7.14) | 2.21 (6.60) | 0.01 (0.01) | 6.21 (8.91)

4. Secondary Outcome: Number of Participants With AEs Due Study Treatment and MIND1 System
Description: Safety and tolerability of the system components was assessed by the device-related AEs, non-serious AEs (NSAEs), serious AEs (SAEs), AEs leading to discontinuation, and unanticipated adverse device effects.
Time Frame: At screening visit (Day -14 to 0), Visit 1 (Day 1) and safety Follow-up (Day 7 [+1] days after the last trial visit)
Population: The Safety sample included all participants who had ingested at least 1 dose of a placebo-embedded IEM, which was the same as the ITT dataset.
Measure: Number; unit: participants
Groups:
- MIND1 System IEM Detection (All Enrolled Participants): On Day 1, for all enrolled participants, a single adhesive patch (paired with the compatible computing device [eg, smartphone] app) was placed on torso (just above the left costal margin, anywhere from the xyphoid to the left mid-axillary line) before the ingestion of the first placebo-embedded IEM tablet. All participants ingested one placebo-embedded IEM tablet approximately every other hour, for a total of 4 ingestions (hours 0, 2, 4, and 6). Placebo-embedded IEM tablets were tested to measure the accuracy of IEM detection by MIND1 system. Clinic staff recorded the time of each ingestion of an IEM. Clinic staff checked the compatible computing device (eg, smartphone) at 30-minute intervals for the presence of a timeline ingestion tile and recorded the time it was detected by the MIND1 system compatible computing device (eg, smartphone).
Arm/Group | MIND1 System IEM Detection (All Enrolled Participants)
Number analyzed (Participants) | 29
participants
  All Treatment-Emergent Adverse Events (TEAEs) | 0
  Treatment-Emergent Serious AEs | 0
  Serious Related TEAEs | 0
  TEAEs led to discontinuation | 0
  Number of death | 0

ADVERSE EVENTS:
Time Frame: At screening visit (Day -14 to 0), Visit 1 (Day 1) and safety Follow-up (Day 7 [+1] days after the last trial visit)
Description: Safety and tolerability was assessed by the frequency and severity of AEs, device-related AEs, SAEs, AEs leading to discontinuation, and unanticipated adverse device effects. Vital signs (heart rate and blood pressure) were analyzed as additional safety variables. The Safety sample included all participants who ingested at least 1 dose of a placebo + IEM, which is the same as the ITT dataset.
Arm/Group | MIND1 System IEM Detection (All Enrolled Participants)
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes